CLINICAL TRIAL: NCT02409043
Title: Neuronal and Glial Biomarkers in Stroke
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201200330
Record Dates: First submitted 2015-02-02; First posted 2015-04-06 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Stroke
Keywords: Stroke; Ischemic stroke; Hemorrhagic stroke; Biomarkers; Angiotensins
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and packed red blood cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control: Non-stroke participants. Blood drawn for analysis of biomarkers.
  Interventions: Other: Blood draw
- Ischemic Stroke: Participants presenting at the University of Florida Shands Emergency Department with an ischemic stroke. Blood drawn at day 1, day 3, and at 2-8 weeks after stroke, NIH stroke scale scores, modified Rankin scale scores, and MRI infarct size assessed in hospital. 3 month modified Rankin scale score collected by phone interview.
  Interventions: Other: Stroke blood draw
- Hemorrhagic Stroke: Participants presenting at the University of Florida Shands Emergency Department with an ischemic stroke. Blood drawn at day 1, day 3, and at 2-8 weeks after stroke, NIH stroke scale scores, modified Rankin scale scores, and MRI infarct size assessed in hospital. 3 month modified Rankin scale score collected by phone interview.
  Interventions: Other: Stroke blood draw
- Stroke Mimic: Participants presenting at the University of Florida Shands Emergency Department with signs and symptoms resembling a stroke, but which are determined to be from another cause. Blood drawn during initial emergency room evaluation.
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — Blood drawn for comparison with other groups
  Groups: Control; Stroke Mimic
Other: Stroke blood draw — Participants presenting at the University of Florida Shands Emergency Department with an ischemic stroke. Blood drawn at day 1, day 3, and at 2-8 weeks after stroke, NIH stroke scale scores, modified Rankin scale scores, blood pressure, MRI infarct volumes, and hospital length of stay taken from the medical records. 3 month modified Rankin scale score collected by phone interview.
  Other Names: Information collection
  Groups: Hemorrhagic Stroke; Ischemic Stroke

SUMMARY:
The purpose of this research study is to determine if there are molecules in the blood that indicate when a person has had a stroke, and what type of stroke they have had, so that appropriate treatment may be begun as soon as possible. This study is also being conducted to determine whether these molecules can help to predict long-term health following stroke. Some of these potential molecules, also called biomarkers, include Neuronal biomarker ubiquitin C-terminal hydrolase-L1 (UCH-L1), Glial markers such as glial fibrillary acidic protein (GFAP), and a neuroprotective enzyme called angiotensin converting enzyme 2 (ACE2), which has activity that has been shown to be helpful cardiovascular disease and shown to be altered in animal models of acute stroke, where it is also shown to provide neuronal protection.

DETAILED DESCRIPTION:
Research Plan Participants will be recruited from those presenting at Shands University of Florida (UF) hospital emergency room within the early hours after symptom onset, during which time a blood draw will be taken. Either in the emergency room, intensive care unit, or general hospital ward, a member of the study team will obtain informed consent for study participation within 24 hours of the first blood draw. The study team will provide the participant or legally authorized representative (LAR) with the consent form to read and will explain the study to the participant or LAR using the consent form as a guide. Time will be given to allow the participant or LAR to read the consent form and any questions will be answered. If the participant or LAR agrees to participate, then the study team member will have the participant sign the consent form and a copy of the signed form will be given for participants' records.

Study procedure: Information will be collected from medical records to determine the type and severity of stroke that the participant had and the time of stroke onset. Three 10cc samples of blood will be drawn from 90 participants with stroke (45 with ischemic stroke and 45 with hemorrhagic stroke). Samples of blood will also be drawn from 45 controls and 45 patients with stroke mimics, clinical symptoms that could be stroke but are determined to be due to another cause (e.g. transient ischemic attack). The first 10cc will be drawn within 18 hours of stroke onset and the second will be drawn 72 hours following stroke onset. The third will be obtained at the UF Neurology outpatient clinic 2-8 weeks after stroke. The first blood sample will be drawn during the initial evaluation in the ER prior to obtaining informed consent. This is due to the hectic ER environment and the need for the participant or LAR to be making serious medical decisions during this initial evaluation; factors which make this a non-ideal time to perform the informed consent process. The blood sample will then be stored using only the de-identified participant number for identification. Once the participant's condition has stabilized and no other serious medical decisions are being made, a study team member will approach the participant or LAR for the informed consent process as described above.

If the informed consent is obtained within 24 hours of obtaining the first blood sample then the participant will be enrolled in the study, the stored blood sample will be kept for further processing, the second and third blood samples will be drawn as previously described and testing for the aforementioned panel of biomarkers will be performed on the blood samples. If the participant or LAR declines to participate in the study or if informed consent is not obtained within 24 hours of the obtaining the first blood sample: 1) the stored blood sample will not be used for any purpose, 2) the stored blood sample will be completely destroyed within 24 hours of knowledge that the participant will not participate in the study and 3) no further blood samples will be obtained. Finally, participant's will be asked to complete a brief (less than 5 minute) phone survey 3 months after stroke to assess long-term stroke disability.

ELIGIBILITY:
Inclusion Criteria:

* Stroke, ischemic or hemorrhagic, is confirmed by clinical and/or imaging evidence
* For control participants, no acute or recent stroke

Exclusion Criteria:

* Onset of stroke symptoms cannot be confirmed to be less than 18 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals experiencing stroke symptoms who present at the University of Florida Shands Emergency Department or non-stroke control participants. These individuals will be invited to participate as study participants by a study representative within the first 24 hours after having a blood draw in the emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Acute Serum ACE2 Activity Levels | Day 1
  Serum and whole blood will be analyzed for levels of ACE2 activity. These markers will be assessed for their value as biomarkers of stroke subtype and long-term outcome.
Subacute Serum ACE2 Activity Levels | Day 3
  Serum and whole blood will be analyzed for levels of ACE2 Activity.
Follow-up Serum ACE2 Activity Levels | 8 weeks
  Serum and whole blood will be analyzed for levels of ACE2 Activity. This last time point will be assessed after discharge from the hospital at the time that the patient returns to the UF Neurology Clinic for their follow-up visit.

SECONDARY OUTCOMES:
Initial NIH Stroke Scale Score | Day 1
  NIH stroke scale scores will obtained as part of the normal care and are scored with points being assigned for neurological deficits (0 = best possible, highest number = best possible) in areas of motor control of the arm (0-4), leg (0-4) sensory perception (0-2), language (0-3), limb ataxia (0-2), gaze (0-2), level of consciousness (0-3), orientation (0-2), response to commands (0-2), facial palsy (0-3), visual (0-3), dysarthria (0-2), and extinction (0-2), and is used to assess the level of neurological deficit from the stroke.
Recovery NIH Stroke Scale Score | Day 14
  NIH stroke scale scores will obtained as part of the normal care and are scored with points being assigned for neurological deficits (0 = best possible, highest number = best possible) in areas of motor control of the arm (0-4), leg (0-4) sensory perception (0-2), language (0-3), limb ataxia (0-2), gaze (0-2), level of consciousness (0-3), orientation (0-2), response to commands (0-2), facial palsy (0-3), visual (0-3), dysarthria (0-2), and extinction (0-2), and is used to assess the level of neurological deficit from the stroke.
Initial infarct size from brain imaging studies | Day 1
  Infarct size will be measured as part of the normal care by MRI volumetric analysis in cm cubed and may range from less than a cm cubed to 20 cm cubed or greater depending on the extent of the stroke. This is meant to assess the size of the stroke.
Recovery infarct size from brain imaging studies | Day 14
  Infarct size will be measured as part of the normal care by MRI volumetric analysis in cm cubed and may range from less than a cm cubed to 20 cm cubed or greater depending on the extent of the stroke. This is meant to assess the size of the stroke.
Initial modified Rankin Score | Day 1
  Initial modified Rankin scale scores will be acquired in hospital as a part of the normal care and by a follow-up phone interview at 3 months. This is scored as follows:
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Recovery modified Rankin Score | Day 14
  Initial modified Rankin scale scores will be acquired in hospital as a part of the normal care and by a follow-up phone interview at 3 months. This is scored as follows:
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Long-term modified Rankin Score | 3 months
  Initial modified Rankin scale scores will be acquired in hospital as a part of the normal care and by a follow-up phone interview at 3 months. This is scored as follows:
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Acute Serum GFAP Levels | Day 1
  Serum and whole blood will be analyzed for levels of GFAP. These markers will be assessed for their value as biomarkers of stroke subtype and long-term outcome.
Subacute Serum GFAP Levels | Day 3
  Serum and whole blood will be analyzed for levels of GFAP. These markers will be assessed for their value as biomarkers of stroke subtype and long-term outcome.
Follow-up Serum GFAP Levels | 8 weeks
  Serum and whole blood will be analyzed for levels of GFAP. These markers will be assessed for their value as biomarkers of stroke subtype and long-term outcome. This last time point will be assessed after discharge from the hospital at the time that the patient returns to the UF Neurology Clinic for their follow-up visit.
Acute Serum UCH-L1 Levels | Day 1
  Serum and whole blood will be analyzed for levels of UCH-L1. These markers will be assessed for their value as biomarkers of stroke subtype and long-term outcome.
Subacute Serum UCH-L1 Levels | Day 3
  Serum and whole blood will be analyzed for levels of UCH-L1. These markers will be assessed for their value as biomarkers of stroke subtype and long-term outcome.
Follow-up Serum UCH-L1 Levels | 8 weeks
  Serum and whole blood will be analyzed for levels of UCH-L1. These markers will be assessed for their value as biomarkers of stroke subtype and long-term outcome. This last time point will be assessed after discharge from the hospital at the time that the patient returns to the UF Neurology Clinic for their follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Harry Nick, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States